CLINICAL TRIAL: NCT01618994
Title: Validation Study for Robotic Surgery Simulator
Status: Completed | Type: Observational
Sponsor: Atlantic Health System (Other)
Collaborators: Intuitive Surgical (Industry)
Responsible Party: Sponsor
Other Study IDs: R11-01-018
Record Dates: First submitted 2012-06-11; First posted 2012-06-14 (Estimated); Last update posted 2017-06-09 (Actual); Status verified 2017-06

CONDITIONS: Pelvic Organ Prolapse
Keywords: Robotic Simulator; EBL; Robotic Surgeons; Intuitive Surgical; simulation modules; benchmarks; Morristown Protocol; Study Surgeons; Control Surgeons; Expert Surgeons; dual-console daVinci system; blinded skill assessment
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Expert Surgeons: Gynecologic robotic surgeons, each averaging >75 robotic cases per year
  Interventions: Procedure: Performing robotic supracervical hysterectomy
- Study Surgeons: Gynecologic surgeons who are completely naive to robotics
  Interventions: Procedure: Performing robotic supracervical hysterectomy
- Control Surgeons: Gynecologic surgeons with full robotic privileges but were not averaging more than 2 cases a month and had never used the simulator
  Interventions: Procedure: Performing robotic supracervical hysterectomy

INTERVENTIONS:
Procedure: Performing robotic supracervical hysterectomy — All groups were recorded, times and graded on their performance during a robotic supracervical hysterectomy

SUMMARY:
A study to determine whether completing a rigorous simulation protocol could provide novice robotic surgeons with actual advanced surgical skills in an operating room setting.

DETAILED DESCRIPTION:
Objective: To determine whether a group of surgeons otherwise naive to robotic techniques could demonstrate proficiency during their first robotic supracervical hysterectomy having only received simulator and pig lab training.

Primary outcome measure: As measured by time spent on the surgeon console from beginning of hysterectomy until the end of cervical amputation.

Secondary Outcome measures:

1. Blood loss- as measured by the blood suctioned into the canister throughout the hysterectomy and at the end of the amputation discounting irrigation volume.
2. Surgical skill rating- All procedures will be recorded and rated by a blinded investigator according to a standardized surgical skills evaluation sheet.
3. Surgeon console biometrics- As measured by controller movements and grips
4. Novice robotic surgeon data: Descriptive Operative data of surgeons who did not participate in robotic simulator training.

Methods: To create the simulator protocol, 5 robotic surgeons (each averaging >75 robotic cases per year) performed all 28 simulation modules available on the da Vinci Skills Simulator. To establish "expert benchmarks", they picked the 10 simulator modules they thought were most beneficial to robotic novices', and they performed each of these 10 modules to the best of their ability >5 times. The data was used to create benchmarks in which all parameters of these 10 modules were taken into account (i.e. not just the time to completion). Thus the "Morristown Protocol" was established- whereby successful completion of the protocol required passing every parameter of all 10 simulator modules at the expert level.

We then recruited community board-certified OB-GYN's who were completely naive to robotics and offered them full robotic training free-of-charge as long as they could pass the "Morristown Protocol" as their very first step in the training process. These "study surgeons" were given 24/7 access to the da Vinci Skills Simulator and simply asked to complete the protocol at their own pace. Within a week of doing so, they went through the standardized Intuitive Surgical pig lab and then performed their first ever robotic surgery- a supracervical hysterectomy- as our main outcome measure. These cases were performed using the dual-console daVinci system with one of the senior authors on the other console ready to step in if necessary.

Two sets of comparative benchmarks for this surgical procedure has been established. Our "expert surgeons" each performed supracervical hysterectomies for the study- as did a group of "control surgeons". These "control surgeons" had full robotic privileges but were not averaging more than 2 cases per month and had never used the simulator. Operative time, EBL, and a blinded skill assessment (of videos) were compared for all cases among the 3 surgeon groups using t-tests.

ELIGIBILITY:
Inclusion Criteria:

* Must not have performed a da Vinci assisted surgery

Exclusion Criteria:

* prior experience on the da Vinci system or the robotic simulator

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Gynecologic surgeons with no robotic experience
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2011-04; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Surgical Time | At end of cervical amputation
  As measured by time spent on the surgeon console from beginning of hysterectomy until the end of cervical amputation

SECONDARY OUTCOMES:
Blood Loss | End of cervical amputation
  As measured by the blood suctioned into the canister throughout the hysterectomy and at the end of the amputation discounting irrigation volume
Surgical Skill Rating | Within a month of the performed surgery
  All procedures will be recorded and rated by a blinded investigator according to a standardized surgical skills evaluation sheet
Surgeon Console Biometrics | during surgery
  As measured by controller movements and grip
Novice Robotic Surgeon Data | Within a month of the performed surgery
  Descriptive Operative data of surgeons who did not participate in robotic simulator training

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Culligan, MD, Principal Investigator — Atlantic Health System; Charbel Salamon, MD, Principal Investigator — Atlantic Health System
Locations (1):
- Morristown Medical Center, Morristown, New Jersey, United States